CLINICAL TRIAL: NCT03521102
Title: An ED-based Randomized Trial of IV Acetaminophen Versus IV Hydromorphone for Elderly Adults With Acute Severe Pain
Brief Title: Acetaminophen Versus IV Hydromorphone for Pain in the Elderly in the ED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-8876
Record Dates: First submitted 2018-04-26; First posted 2018-05-11 (Actual); Results first posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Acetaminophen; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Acetaminophen 1000mg IV (Experimental): NRS pain score will be obtained at baseline, 15, 30, 45, 60, 90, 120, and 180 minutes following completion of intervention. Adverse events will be recorded every 15 minutes for the duration of the study protocol. Participants will be reassessed for the need of additional pain control at 60 minutes.
  Interventions: Drug: Acetaminophen 1000mg IV
- Hydromorphone 0.5mg IV (Active Comparator): NRS pain score will be checked at 5 minutes and every 15 minutes thereafter for 120 minutes. Adverse events will be recorded every 15 minutes for the duration of the study protocol. The need for additional pain control will be assessed at 60 minutes.
  Interventions: Drug: Hydromorphone 0.5 mg IV

INTERVENTIONS:
Drug: Acetaminophen 1000mg IV — 1000mg of IV acetaminophen in 100ml of normal saline, administered as an intravenous drip over 10 minutes + 2ml of normal saline, administered as a slow intravenous push
  Arms: Acetaminophen 1000mg IV
Drug: Hydromorphone 0.5 mg IV — 100ml of normal saline, administered as an intravenous drip over 10 minutes, + 0.5mg of IV hydromorphone in 2ml of normal saline, administered as a slow intravenous push
  Arms: Hydromorphone 0.5mg IV

SUMMARY:
Intravenous opioids are the mainstay of acute, severe pain treatment in Emergency Departments (ED) across the country. Acetaminophen, given orally, has also been used for treatment of mild to moderate pain. The more potent intravenous (IV) form of acetaminophen has been widely used in Europe for more than 20 years as post-surgical analgesia and received full FDA approval in the USA in 2010. As part of a continuing set of studies whose goal is to optimize treatment of pain among elderly ED patients, this randomized study will compare efficacy and safety of IV acetaminophen to IV hydromorphone.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal to 65 or greater
2. Pain onset within 7 days with severe pain
3. Has capacity to provide informed consent
4. Understanding English or Spanish

Exclusion Criteria:

1. Use of tramadol or opioids within 7 days
2. Use of acetaminophen or non-steroidal anti-inflammatory medications within 8 hours
3. Chronic pain syndrome: daily pain for > 3 months. Sickle cell anemia, osteoarthritis, fibromyalgia, and peripheral neuropathies
4. Conditions which may affect acetaminophen or opioid metabolism such as cirrhosis (Child Pugh A or worse), kidney impairment (CKD 3 or worse), active hepatic disease or severe dehydration
5. Alcohol intoxication
6. Systolic blood pressure: < 100 mmHg
7. Heart rate: < 60 beats per minute
8. Oxygen saturation: < 95% on room air
9. Use of monoamine oxidase (MAO) inhibitors in the past 30 days
10. Use of transdermal pain patch or oral opioid > 10 days in the prior month
11. Prior enrollment in the same study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 162 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Friedman, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kolli S, Friedman BW, Latev A, Chang AK, Naeem F, Feliciano C, Afrifa F, Walker C, Izzo A, Irizarry E. A Randomized Study of Intravenous Hydromorphone Versus Intravenous Acetaminophen for Older Adult Patients with Acute Severe Pain. Ann Emerg Med. 2022 Nov;80(5):432-439. doi: 10.1016/j.annemergmed.2022.06.016. Epub 2022 Aug 12. PMID 35965162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in August 2018, paused between March and June 2020, and concluded in October 2021. A total of 2,363 patients were screened for participation of which 162 were enrolled from two urban emergency departments in Bronx, NY.
Groups:
- Hydromorphone 0.5mg IV: Hydromorphone 0.5 mg IV: 100ml of normal saline, administered as an intravenous drip over 10 minutes, + 0.5mg of IV hydromorphone in solution with 2mL of normal saline, administered as a slow intravenous push.
Period: Overall Study
Arm/Group | Acetaminophen 1000mg IV | Hydromorphone 0.5mg IV
Started | 81 | 81
Completed | 81 | 81
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen 1000mg IV | Hydromorphone 0.5mg IV | Total
Number analyzed (Participants) | 81 | 81 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (8) | 74 (6) | 75 (7)
Age, Customized [Count of Participants; unit: Participants]
  60-69 years old | 23 | 22 | 45
  70-79 years old | 40 | 45 | 85
  80-89 years old | 12 | 14 | 26
  >=90 years old | 6 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 51 | 107
  Male | 25 | 30 | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 81 | 81 | 162
Duration of Pain [Median (Inter-Quartile Range); unit: Minutes] | 2 [1 to 4] | 2 [1 to 3] | 2 [1 to 4]
NRS Pain Score (0-10) [Median (Inter-Quartile Range); unit: score on a scale] — Pain intensity was assessed at baseline using an NRS (numeric rating scale) to assess participants' pain on a linear range of 0-10. Participants were asked to verbalize level of pain on a scale where 0 represented "no pain" and 10 represented "the worst pain imaginable." As such, a higher NRS baseline pain score denoted a higher degree of pain being felt prior to treatment.
  score on a scale | 10 [8 to 10] | 10 [8 to 10] | 10 [8 to 10]
Location of Pain [Count of Participants; unit: Participants]
  Abdomen/Flank/Pelvis | 52 | 55 | 107
  Back/Neck | 6 | 7 | 13
  Chest | 1 | 6 | 7
  Extremity | 21 | 11 | 32
  Head | 0 | 2 | 2
  Widespread | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement in NRS Pain Score
Description: Pain improvement was assessed using an NRS (numeric rating scale) to assess pain on a range of 0-10. Participants were asked to verbalize intensity of pain on the scale with zero meaning "no pain" and 10 meaning "the worst pain imaginable." Pain was assessed at baseline and 60 minutes later to determine if clinically important improvement in pain was achieved. Clinically important improvement in pain was defined as an improvement of >=1.3 points on the 0-10 scale.
Time Frame: 60 minutes following administration of medication
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen 1000mg IV | Hydromorphone 0.5mg IV
Number analyzed (Participants) | 81 | 81
Participants | 62 | 63

2. Secondary Outcome: Need for Rescue Medication
Description: Number of participants who required additional analgesic medication for the treatment of pain at any time during their ED course.
Time Frame: 120 minutes following administration of medication
Population: Study participants did not receive any additional medication before the assessment of the primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen 1000mg IV | Hydromorphone 0.5mg IV
Number analyzed (Participants) | 81 | 81
Participants | 37 | 31

3. Secondary Outcome: Improvement in NPS Pain Score by >=50%
Description: The number of patients who minimally achieved a 50% improvement in NPS pain score from 0 to 60 minutes.
Time Frame: 60 minutes after administration of medication
Population: Study participants did not receive any additional medication before the assessment of the primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen 1000mg IV | Hydromorphone 0.5mg IV
Number analyzed (Participants) | 81 | 81
Participants | 30 | 43

ADVERSE EVENTS:
Time Frame: Participants were queried for the emergence of new symptoms after receipt of the investigational medication. Affirmative responses were followed with an open-ended question eliciting details regarding side effects 30 and 60 minutes after medication administration.
Arm/Group | Acetaminophen 1000mg IV | Hydromorphone 0.5mg IV
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/81
Other Adverse Events (participants affected / at risk) | 6/81 | 10/81
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetaminophen 1000mg IV (N=81) | Hydromorphone 0.5mg IV (N=81)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4)
Drowsiness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Discomfort NEC (General disorders) | 1 (1) | 1 (1) — NEC - not elsewhere classified

LIMITATIONS AND CAVEATS:
Enrollment limited to 2 urban EDs, excluding a large number of patients who had been screened. Results may not be generalizable to all older patients with acute severe pain Dose ranging studies were not conducted to help optimize hydromorphone dosage An arbitrary value (1.3) was selected as the minimum clinically important improvement threshold The study relied on the clinical attending physician's judgment of whether opioids were indicated. Would not account for local practices

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT03521102/Prot_SAP_001.pdf